CLINICAL TRIAL: NCT06422884
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Controlled Trial Evaluating the Safety and Efficacy of ENV-101 in Patients With Lung Fibrosis (WHISTLE-PF Trial)
Brief Title: A Phase 2 Trial of ENV-101 in Patients With Lung Fibrosis (WHISTLE-PF Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Biomedicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENV-IPF-103
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis; Progressive Fibrosing Interstitial Lung Disease
Keywords: taladegib; hedgehog pathway inhibitor; pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — LY2940680

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ENV-101 Low Dose (IPF Population) (Experimental)
  Interventions: Drug: ENV-101
- ENV-101 Mid Dose (IPF Population) (Experimental)
  Interventions: Drug: ENV-101
- ENV-101 High Dose (IPF Population) (Experimental)
  Interventions: Drug: ENV-101
- Placebo (IPF Population) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENV-101 — oral tablet, dosed once a day
  Other Names: taladegib
  Arms: ENV-101 High Dose (IPF Population); ENV-101 Low Dose (IPF Population); ENV-101 Mid Dose (IPF Population)
Drug: Placebo — oral tablet, dosed once a day
  Arms: Placebo (IPF Population)

SUMMARY:
The goal of this clinical trial is to evaluate the impact that ENV-101 has on lung function and key measures of fibrosis in adult patients with idiopathic pulmonary fibrosis (IPF). Another goal of this study is to better understand the safety and tolerability of ENV-101 in this patient population.

DETAILED DESCRIPTION:
This trial is a 6-month, randomized, double-blind, controlled, dose-ranging trial of ENV-101 in adult patients with idiopathic pulmonary fibrosis (IPF). Patients are allowed to continue treatment with approved standard of care (e.g., nintedanib, pirfenidone) during the trial. Patients will be randomized to one of 3 dose levels of ENV-101 or placebo at baseline. The objectives of this trial are to characterize the efficacy, antifibrotic activity, and safety of ENV-101 to select the Phase 3 dose of ENV-101.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 40 years old with an IPF diagnosis as confirmed by the Investigator.
* Percent predicted FVC of ≥ 45% at study start.
* Percent predicted diffusing capacity of lung for carbon monoxide (DLCO) ≥ 25%, adjusted for hemoglobin (Hgb) at study start.
* Ability to perform spirometry tests.
* Either stable treatment with standard of care (SoC) [i.e., antifibrotics, immunosuppressants (PPF only)] for at least 3 months prior to study start or not treated with SoC for at least 8 weeks prior to study start.

Exclusion Criteria:

* Evidence of other known causes of interstitial lung disease (ILD).
* Forced expiratory volume in one second (FEV1)/FVC ratio <0.7 at study start.
* History of malignancy, including carcinoma during the preceding 5 years from study start, with the following exceptions:

  1. Prior history of in situ melanoma, basal or squamous cell skin cancer if treated with curative therapy.
  2. Patients with prostate cancer that are managed by surveillance.
  3. Patients with ductal carcinoma in situ, treated surgically with curative intent.
* Patients with moderate to severe hepatic impairment (Child-Pugh B and C).
* Smoking (including vaping) within 6 months of study start; current smoker, or unwillingness to refrain from smoking during the clinical trial duration.
* Active or suspected alcohol or drug abuse in the opinion of the Investigator.
* Currently enrolled in another investigational device or drug trial, or less than 3 months from study start since ending another investigational device or drug trial(s) or receiving other investigational treatment(s).
* Presence of active infection at study start or confirmed active human immunodeficiency virus (HIV), Hepatitis B virus (HBV) or Hepatitis C virus (HCV).
* Major surgery requiring hospitalization (according to the Investigator) performed within 3 months prior to study start or planned during the course of the trial. Being on a transplant list is allowed.
* Occurrence of serious illness requiring hospitalization within 90 days prior to study start.
* Current or previous use (within 28 days prior to study start) of the following:

  1. Endothelin receptor antagonist
  2. Riociguat
  3. Prostacyclin or prostacyclin analogue
  4. Radiation to the lungs
  5. Oral corticosteroids >15 mg/day
* Use of cyclophosphamide or tocilizumab within 8 weeks, or rituximab within 6 months, prior to study start.
* Use of drugs that are known moderate or stronger CYP3A4 inhibitors or inducers within 14 days prior to study start. Patients must also agree not to eat fruits that inhibit CYP3A4 such as grapefruit, Seville oranges, pomelo and star fruit.
* Patients of reproductive potential who are sexually active and unwilling to use birth control for the duration of the study and for 3 months after their final dose of study drug.
* Females that are pregnant or nursing.
* Patients that are unwilling to refrain from blood or blood product donation for the duration of the study and for 30 days after their final dose of study drug.
* Males who are unwilling to refrain from sperm donation and females who are unwilling to refrain from egg donation for the duration of the study and for 3 months after their final dose of study drug.
* Patients with a history of a severe allergic reaction or anaphylactic reaction or known hypersensitivity to any component of ENV-101.
* Patients who have previously taken ENV-101.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rate of change in percent predicted forced vital capacity (ppFVC) compared to placebo | Baseline and Week 24
  ppFVC is a measure of lung function

SECONDARY OUTCOMES:
Absolute change in FVC (mL) compared to placebo | Baseline and Week 24
  FVC is a measure of lung function
Time to disease progression (absolute decline in ppFVC >10%, IPF-related hospitalization, or death) compared to placebo | Baseline and Week 24
Absolute change in the Living with Pulmonary Fibrosis Symptoms (L-PF Symptoms) Questionnaire Cough domain score compared to placebo | Baseline and Week 24
  The L-PF Symptoms Questionnaire Cough domain consists of 6 questions regarding a subject's experience with cough over the prior 24 hours. Questions have response options on a five-point numeric rating scale with an anchor of 0 ("Not at all") to 4 ("Extremely"). Total score for the Cough domain is normalized to the range 0 to 100, with higher scores indicating greater impairment.
Absolute change in the L-PF Symptoms Questionnaire Dyspnea domain score compared to placebo | Baseline and Week 24
  The L-PF Symptoms Questionnaire Dyspnea domain consists of 12 questions regarding a subject's experience with dyspnea (shortness of breath) over the prior 24 hours. Questions have response options on a five-point numeric rating scale with an anchor of 0 ("Not at all") to 4 ("Extremely"). Total score for the Dyspnea domain is normalized to the range 0 to 100, with higher scores indicating greater impairment.
Absolute change in the L-PF Symptoms Questionnaire Fatigue domain score compared to placebo | Baseline and Week 24
  The L-PF Symptoms Questionnaire Fatigue domain consists of 5 questions regarding a subject's experience with fatigue over the prior 24 hours. Questions have response options on a five-point numeric rating scale with an anchor of 0 ("Not at all") to 4 ("Extremely"). Total score for the Fatigue domain is normalized to the range 0 to 100, with higher scores indicating greater impairment.
Absolute change in total lung capacity (TLC) by chest high-resolution computed tomography (HRCT) imaging compared to placebo | Baseline and Week 24
  HRCT is a method of imaging which is more precise than chest x-ray in the diagnosis and monitoring of diseases of the lung tissue and the airways.
Absolute change in % quantitative interstitial lung disease (QILD) by chest HRCT imaging compared to placebo compared to placebo | Baseline and Week 24
Absolute change in % quantitative ground glass opacity (QGG) by chest HRCT imaging compared to placebo | Baseline and Week 24
Absolute change in % quantitative lung fibrosis (QLF) by chest HRCT imaging compared to placebo | Baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lancaster, M.D., Study Director — Endeavor Biomedicines
Locations (72):
- Argentina (3):
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Buenos Aires
  - Research Site, Mendoza
- Australia (8):
  - Research Site, Camperdown, New South Wales
  - Research Site, Macquarie Park, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, South Brisbane, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Nedlands, Western Australia
- Austria (2):
  - Research Site, Graz, Styria
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Dinant, Namur
  - Research Site, Brussels
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Trois-Rivières, Quebec
- France (9):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Tours
- Germany (6):
  - Research Site, Giessen, Hesse
  - Research Site, Immenhausen, Hesse
  - Research Site, Hanover, Lower Saxony
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Berlin
  - Research Site, Leipzig
- Ireland (3):
  - Research Site, Dublin, Leinster
  - Research Site, Cork, Munster
  - Research Site, Dublin
- Italy (6):
  - Research Site, Bologna, Forli-Cesena
  - Research Site, Padua, Padua
  - Research Site, Florence, Tuscany
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Turin
- Research Site, Kuala Lumpur, Selangor, Malaysia
- Mexico (7):
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Nicolás de los Garza, Nuevo León
  - Research Site, San Juan del Río, Querétaro
  - Research Site, Chihuahua City
  - Research Site, Mexico City
  - Research Site, Oaxaca City
  - Research Site, Puebla City
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Hamilton
- South Korea (8):
  - Research Site, Seoul, (Deogyang District)
  - Research Site, Ulsan, (Dong District)
  - Research Site, Seoul, (Gangnam District)
  - Research Site, Busan, (Haeundae District)
  - Research Site, Seoul, (Seongbuk District)
  - Research Site, Seoul, (Songpa District)
  - Research Site, Seoul, (Yongsan District)
  - Research Site, Seoul
- United Kingdom (8):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, Exeter
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Londonderry

IPD SHARING:
Plan to Share IPD: No